CLINICAL TRIAL: NCT05170971
Title: The Clinical Efficacy and Safety of Fecal Microbiota Transplantation in Patients With Acute-on-chronic Liver Failure
Brief Title: Fecal Microbiota Transplantation for Liver Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Principal Investigator, xulanman, Head of Infection Department, Ningbo Medical Center Lihuili Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KJ2019PJ021
Record Dates: First submitted 2021-05-27; First posted 2021-12-28 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Liver Failure
Keywords: fecal microbiota transplantation; gut-liver axis; liver failure
MeSH Terms: conditions — Liver Failure | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fecal microbiota transplantation (Other): The fecal bacteria were transplanted once every 5 days for a total of 4 times.
  Interventions: Other: fecal microbiota transplantation

INTERVENTIONS:
Other: fecal microbiota transplantation — The fecal bacteria were transplanted once every 5 days for a total of 4 times

SUMMARY:
To investigate the safety, adverse reactions and therapeutic effects of fecal microbiota transplantation on patients with liver failure;to investigate the effect of fecal microbiota transplantation on the intestinal microecology and "gut-liver axis immune system" of liver failure, and further optimization of fecal microbiota transplantation technology.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign informed consent
* Patients aged 18-65
* According to the diagnosis standard of liver failure in the guide for diagnosis and treatment of liver failure (2018 Edition), the eligible patients are included, that is, on the basis of chronic liver disease, the syndrome with acute jaundice deepening and coagulation dysfunction as the manifestation of liver failure caused by various inducements can be combined with complications such as Hepatoencephalopathy, ascites, electrolyte disorder, infection, hepatorenal syndrome, hepatopulmonary syndrome, etc And extrahepatic organ failure. The patient's jaundice deepened rapidly, the serum TBIL ≥ 10 × ULN or the daily rise ≥ 17.1 μ mol / L; there was bleeding, PTA ≤ 40% (or INR ≥ 1.5)

Exclusion Criteria:

* Patients with severe heart failure, COPD, cerebrovascular accident, nephrotic syndrome, etc;
* Patients with gastrointestinal bleeding, pulmonary infection, septicemia, etc
* Patients with liver cancer, lung cancer, lymphoma and other malignant tumors
* Patients taking anticoagulants, mental diseases and immune diseases for a long time
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver function change | Blood samples were collected 1 week before faecal bacteria transplantation, and followed up at 5 day, 10 day, 15 day, 20 day, 4 and 8 weeks after faecal bacteria transplantation, respectively
  The investigators need to monitor the changes in liver and kidney function before and after faecal bacteria transplantation，such as ALT、AST、GGT 、TBIL(The units of these indices are U/L).
Coagulation function change | Blood samples were collected 1 week before faecal bacteria transplantation, and followed up at 5 day, 10 day, 15 day, 20 day, 4 and 8 weeks after faecal bacteria transplantation, respectively
  Prothrombin activity are one of the indexes to evaluate the degree of liver failure in patients.The units of this indices is %.
Model for end-stage liver disease score change | Model for end-stage liver disease score were obtained separately in 1 week before faecal bacteria transplantation, and to access once again at 5 day, 10 day, 15 day, 20 day, 4 and 8 weeks after faecal bacteria transplantation, respectively
  The model for end-stage liver disease (MELD) score is a prospectively developed and validated scale for the severity of end-stage liver disease.The higher the MELD score, the more severe the liver disease and the greater the risk of death. The fatality rate of patients with MELD between 20 and 30 was more than 30%, that of patients with MELD between 30 and 40 was more than 50%, and that of patients with MELD >40 was more than 70%.
gut microbiota change | Fecal samples were collected 1 week before faecal bacteria transplantation, and change from at 5 day, 10 day, 15 day, 20 day, 4 and 8 weeks after faecal bacteria transplantation, respectively
  Gene sequencing and metabonomics analysis of fecal flora.
Observe the clinical manifestations, safety and adverse reactions of the patients | These indicators were collected 1 week before faecal bacteria transplantation, and change from at 5 day, 10 day, 15 day, 20 day, 4 and 8 weeks after faecal bacteria transplantation, respectively
  Safety and adverse events were assessed including fever, diarrhea and elevated inflammatory markers (such as C-reactive protein and procalcitonin) before and after faecal bacteria transplantation.
proinflammatory cytokine change | Blood samples were collected 1 week before faecal bacteria transplantation, and followed up at 5 day, 10 day, 15 day, 20 day, 4 and 8 weeks after faecal bacteria transplantation, respectively
  IL-17,IL-6,TNF-α, TGF-β, IFN-γ and other cytokines were detected by ELISA(The units of these indices are pg/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Medical Center Lihuili Hospital,Affiliated Lihuili hospital of Ningbo University, Ningbo, Zhejiang, China